CLINICAL TRIAL: NCT04057885
Title: A PILOT STUDY: To Determine the Gait and Functional Improvement in Total Knee Arthroplasty With Use of Orthosensor™ VERASENSE™ Knee System for Soft Tissue Balancing.
Brief Title: To Determine the Gait and Functional Improvement in Total Knee Arthroplasty
Acronym: Orthosensor
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lead Investigator no longer with institution
Sponsor: LifeBridge Health (Other)
Collaborators: Orthosensor, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Orthosensor 101
Record Dates: First submitted 2015-06-12; First posted 2019-08-15 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2019-08

CONDITIONS: Degenerative Arthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Device Arm (Experimental): A prospective series of 10 patients will receive sensor-guided TKA using the this special Orthosensor™ VERASENSE™ Knee System assisted surgery for optimization of soft tissue balance
  Interventions: Device: Orthosensor™ VERASENSE™ Knee System
- Standard of Care (Active Comparator): 10 patients will receive standard of care. Prior to cementing final implants, VERASENSE will be utilized with the standard of care group with the surgeon blinded to the data.
  Interventions: Device: Orthosensor™ VERASENSE™ Knee System

INTERVENTIONS:
Device: Orthosensor™ VERASENSE™ Knee System — A group of patients will receive a total knee arthroplasty using the Orthosensor device

SUMMARY:
This is an observational study to understand the effects of soft-tissue balancing on gait, function and rehabilitation potential after sensor-assisted Total Knee Arthroplasty

DETAILED DESCRIPTION:
The primary objectives of this study are to understand the effects of soft-tissue balancing on Gait, function and rehabilitation potential after sensor-assisted Total Knee Arthroplasty and to correlate Intra-operative subjective feel with OrthoSensor Outputs

Secondary objectives are to quantify and observe pain medication use, swelling, muscle strength and girth, gait efficiency, patient satisfaction, activity levels, functional return (i.e., back to work, resume normal activities) and patient perception of a balanced knee

ELIGIBILITY:
Inclusion Criteria:

* Subject must be a candidate for a primary PCL retaining total knee arthroplasty
* Subject must be diagnosed with one or more of the following conditions:

  1. osteoarthritis
  2. avascular necrosis
  3. rheumatoid or other inflammatory arthritis
  4. post-traumatic arthritis Minimum age: 45 Maximum age: 80
* Subject is likely to be available for all study visits
* Subject is able and willing to sign the informed consent and follow study procedures

Exclusion Criteria

1. Prior total knee arthroplasty
2. ligament insufficiencies
3. prior surgeries such as:

   1. ACL or PCL reconstructions
   2. posterolateral reconstructions
   3. osteotomies
   4. tibia plateau fractures
   5. Range of Motion less than 90 degrees f ) flexion contracture of more than 20 degrees

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with improvement in gait. | 18 months
Proportion of patients not requiring long term rehabilitation. | 18 months
Proportion of patients with improved function as measured by standardized knee scores. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Mont, M.D., Principal Investigator — Director, Rubin Institute for Advanced Orthopedics and Joint Preservation
Locations (1):
- Sinai Hospital of Baltimore, Baltimore, Maryland, United States